CLINICAL TRIAL: NCT03908320
Title: Testing the Feasibility of a Novel Smoking Cessation Intervention by Timing Quit Dates to Menstrual Phase in a Quitline Setting
Brief Title: Menstrual Phase and Smoking Cessation at a State Quitline
Acronym: Project Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Alicia Allen, PhD, MPH, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1805561891
Record Dates: First submitted 2019-03-28; First posted 2019-04-09 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Menstrual Cycle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menstrual Cycle Timing (Experimental)
  Interventions: Other: Menstrual Cycle Timing; Drug: NRT Patch; Behavioral: Cessation Counseling
- Menstrual Cycle Monitoring (Active Comparator)
  Interventions: Other: Menstrual Cycle Timing; Drug: NRT Patch; Behavioral: Cessation Counseling

INTERVENTIONS:
Other: Menstrual Cycle Timing — Quit date is set to menstrual phase.
  Arms: Menstrual Cycle Timing
Other: Menstrual Cycle Timing — Menstrual cycle timing of quit date is monitored
  Arms: Menstrual Cycle Monitoring
Drug: NRT Patch — NRT patch is provided
Behavioral: Cessation Counseling — Cessation counseling is provided

SUMMARY:
Quitlines are efficient and cost-effective treatments for smoking cessation, yet little research has explored how to personalize and optimize quitline services for women. The goal of this project is to explore the feasibility and preliminary efficacy of a quitline intervention that considers the menstrual cycle as compared to standard care for cessation. If funded, the results of this study will directly inform future research on quitline smoking cessation interventions for premenopausal women, including a full scale clinical trial.

DETAILED DESCRIPTION:
Although more than 75% of women who smoke want to quit, they do not have the same success that men have. This is of particular concern as premenopausal women smokers are more likely to experience smoking-related morbidity and mortality than men smokers. Further, mothers are the primary source of secondhand smoke exposure in children. Quitlines are broad reaching, cost-effective programs that disseminate smoking cessation treatment; however, little research has focused on tailoring quitline programs for women. The goal of this study is to investigate how the quit interventions can be informed by the menstrual cycle to improve cessation outcomes in women. This study will enroll 116 women between 18-40 years of age from the Arizona Smokers' Helpline. Menstrual phase identification will be determined using methods from published recommendations. Consistent with existing quitline protocols, participants will receive 4-weeks of NRT (patch) concurrent with six-weeks of telephone-based behavioral coaching. Data will be collected at Baseline, Week 0 (quit day), Week 1, Week 4 (end of treatment), and a follow-up at Month 3 using telephone interviews, validated questionnaires, and dried blood spots (to measure sex hormones to verify menstrual phase and cotinine to verify smoking status). Primary outcomes include determining acceptability and feasibility of this menstrual-cycle based intervention (recruitment and retention rate, the ability to correctly identify the menstrual phase, and overall participant study satisfaction). Smoking cessation outcomes (self-report and/or biochemically verified) will be assessed at Week 1, Week 4 (end of treatment), and at Month 3 follow-up. Finally, we will explore menstrual phase differences in theoretically-relevant factors known to be associated with smoking cessation (e.g., social support, weight concerns, urge coping). Study results will guide protocol development and generate hypotheses for larger-scaled randomized controlled trials. This study is novel and pragmatic, integrating emerging evidence for the role of menstrual-cycle timed quit dates with state-of-the-science quitline cessation programs. If successful, this model can be cost-effectively replicated within state and national quitline programs. It can address the unique barriers to smoking behavior change among premenopausal women, increase successful quit outcomes and reduce disease risk associated with high tobacco-related morbidity rates.

ELIGIBILITY:
Inclusion Criteria:

* Regular smoking
* Regular, natural menstrual cycles
* Interested in quitting

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Contraindications to NRT patch

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility | Week -3
  Average number of participants enrolled per month
Treatment Retention Feasibility | Week 4
  Total number of participants who complete to end of treatment
Follow-up Retention Feasibility | Month 3
  Total number of participants who complete follow-up
Feasibility Menstrual Phase Identification | Week 0
  Total proportion of active participants who have a progesterone level of <2 ng/ml on quit date

SECONDARY OUTCOMES:
Smoking Cessation | Week 4, Month 3
  Biochemically confirmed abstinence
Smoking Cessation | 24 hours, Week 1
  Self-reported abstinence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Pending

REFERENCES:
- [Derived] Chalke AM, Linde-Krieger LB, Allen AM, Nair US. Urge Coping Mediates the Relationship Between Physical Activity and Smoking Outcomes in a Sample of Premenopausal Women Intending to Quit Smoking. Nicotine Tob Res. 2025 Oct 22;27(11):2086-2096. doi: 10.1093/ntr/ntaf081. PMID 40214198